CLINICAL TRIAL: NCT06145243
Title: Comparison of the Effectiveness of Supervised, Video-based and Home-based Resistance Exercise Program in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, Asistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATADEK 2023-10/342
Record Dates: First submitted 2023-11-16; First posted 2023-11-24 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Visual brochure based resistive home exercise group, (Active Comparator): In the 8-week exercise training, the exercise resistance of the patients will start with 60-70% according to1 Repetition Maximum in the first 4 weeks and will be increased to 70-80% according to 1 Repetition Maximum in the last 4 weeks according to the American College of Sports Medicine safe exercise intensity guideline for elderly individuals.
  Interventions: Other: Home based exercise
- Video-based resistive home exercise group (Active Comparator): In the 8-week exercise training, the exercise resistance of the patients will start with 60-70% according to 1 Repetition Maximum in the first 4 weeks and will be increased to 70-80% according to 1 1 Repetition Maximum in the last 4 weeks according to the American College of Sports Medicine safe exercise intensity guideline for elderly individuals.
  Interventions: Other: Video-based resistive exercise
- Supervised resistance exercise group (Experimental): In the 8-week exercise training, the exercise resistance of the patients will start with 60-70% according to 1 Repetition Maximum in the first 4 weeks and will be increased to 70-80% according to 1 Repetition Maximum in the last 4 weeks according to the American College of Sports Medicine safe exercise intensity guideline for elderly individuals.
  Interventions: Other: Supervised resistive exercise

INTERVENTIONS:
Other: Home based exercise — Patients will be given a visual brochure with pictures explaining the exercises. Patients will perform the resistance exercises in the given exercise program for 8 weeks, 2 days a week for 8-12 repetitions and 3 sets using resistance bands.Progress of the home exercise group will be checked by phone every week.
  Arms: Visual brochure based resistive home exercise group,
Other: Video-based resistive exercise — A video recording of the exercises will be taken and given to the patients as a video recording.Patients will perform the resistance exercises in the given exercise program for 8 weeks, 2 days a week for 8-12 repetitions and 3 sets using resistance bands.Progress of the video-based exercise group will be checked by phone every week.
  Arms: Video-based resistive home exercise group
Other: Supervised resistive exercise — Patients will perform their exercises under the supervision of a physiotherapist.Patients will perform the resistance exercises in the given exercise program for 8 weeks, 2 days a week for 8-12 repetitions and 3 sets using resistance bands.
  Arms: Supervised resistance exercise group

SUMMARY:
The aim of this study was to compare the effects of video-based application method of resistance exercise training and supervised exercise training on mobility, body composition, quality of life, fatigue, muscle strength and physical performance in patients with prostate cancer receiving androgen deprivation therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer with at least 1 year of Androgen deprivation therapy treatment
* 65 years of age or older
* No speech and hearing problems

Exclusion Criteria:

* Presence of metastatic cancer focus
* Carrying a pacemaker
* Mental and coordination problems
* Patients with neurological or orthopedic pathology that would prevent participation in exercise

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 8 weeks
  Muscle strength of the patients' reference muscles gluteus maximus, quadriceps, hamstring, gastrocsoleus, gluteus medius, will be evaluated with Hand Held dynamometer.For each muscle group, 3 measurements will be made at 1 minute intervals and the average of the measurements will be accepted as the evaluation result.
Body composition- fat percentage | 8 weeks
  Total body fat percentage, will be measured using Dual-Energy Xray Absorptiometry (DEXA) at baseline and after treatment in percentile.
Body composition- Body mass index( BMI in kg/m^2) | 8 weeks
  Total body fat mass, will be measured using Dual-Energy Xray Absorptiometry (DEXA) at baseline and after treatment in BMI in kg/m^2.
Short Physical Performance Battery | 8 weeks
  The physical performance level of the patients will be assessed with the short physical performance battery, which is a combined test that includes a chair stand test along with gait speed and balance assessment. The maximum score is 12 and a score of ≤8 indicates poor physical performance.
Quality of Life- Functional Assessment of Cancer Therapy - Prostate cancer (FACT-P) | 8 weeks
  FACT-P is a scale that assesses the quality of life of patients with prostate cancer. The 27-question general version consists of sections assessing emotional, social or family, physical and functional status. There are 12 questions about the treatment of patients with prostate cancer and additional concerns. The lowest score is 0 and the highest score is 156. A high score indicates good quality of life.

SECONDARY OUTCOMES:
Grip strength | 8 weeks
  Grip strength was evaluated by hand grip dynamometry. Measurements were performed in affected side according to positions defined by American Society of Hand Therapists (sitting with the shoulder adducted to the side and the elbow flexed 90° with the forearm and wrist in the neutral mid-position)
Fatigue -Functional assessment of chronic illness therapy - fatigue | 8 weeks
  FACIT-F consists of 13 questions assessing the level of fatigue during daily activities in the last week. The maximum score is 52. A high score indicates a high level of fatigue. It is a Likert-type scale scored between 0-4.
Sarcopenia Risk Survey | 8 weeks
  Sarcopenia Risk Survey is a 5-item questionnaire self-reported by patients as a screening for sarcopenia risk. It assesses 5 components: strength, supported walking, getting up from a chair, climbing stairs and falling. Scoring for each component ranges from 0-2, with a total score of 0-10. A score of 4 or more indicates sarcopenia.
Anxiety - The Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) Anxiety and depression levels of the patients will be evaluated with the HADS questionnaire.This scale has subscales for anxiety and depression. It includes a total of 14 questions. Seven items measure anxiety and the other seven items measure depression. The lowest score is "0" and the highest score is "21". An increase in the total score indicates an increase in the level of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Cemil Taşcıoğlu Training and Research Hospital, Istanbul, Turkey (Türkiye)